CLINICAL TRIAL: NCT06221150
Title: Ultrasound-guided Bilateral Two Levels Serratus Anterior Plane Block in Pediatric Cardiac Surgery With Median Sternotomy : A Randomized Controlled Trial
Brief Title: Bilateral Two Levels Serratus Anterior Plane Block in Pediatric Cardiac Surgery With Median Sternotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Madkour, Associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MD-341-2023
Record Dates: First submitted 2024-01-05; First posted 2024-01-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-01

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAPB group (Experimental): bilateral two-level SAPB is performed with the guidance of ultrasound. While the patient is in the supine position with their arms abducted, the US probe is placed in longitudinal plane to visualize and count the ribs down from the clavicle while moving the transducer laterally and distally to identify the muscles overlying the 3rd and 6th ribs at the mid axillary line. Using in- plane approach, a 22-gauge short bevel needle is inserted and advanced to the plane deep to the serratus anterior muscle at the level of 3rd and 6th ribs bilaterally in succession over which a total volume of 1.5ml/kg bupivacaine 0.125% is divided and injected (0.75ml/kg on each side); with total dose not exceeding 2.5 mg/kg.
  Interventions: Procedure: Bilateral two level serratus anterior block
- control group (No Intervention): Intraoperative fentanyl without nerve block

INTERVENTIONS:
Procedure: Bilateral two level serratus anterior block — bilateral two-level SAPB is performed with the guidance of ultrasound. While the patient is in the supine position with their arms abducted, the US probe is placed in longitudinal plane to visualize and count the ribs down from the clavicle while moving the transducer laterally and distally to identify the muscles overlying the 3rd and 6th ribs at the mid axillary line. Using in- plane approach, a 22-gauge short bevel needle is inserted and advanced to the plane deep to the serratus anterior muscle at the level of 3rd and 6th ribs bilaterally in succession over which a total volume of 1.5ml/kg bupivacaine 0.125% is divided and injected (0.75ml/kg on each side); with total dose not exceeding 2.5 mg/kg.
  Other Names: Bilateral SAPB
  Arms: SAPB group

SUMMARY:
The serratus anterior plane block (SAPB) is an anterolateral thoracic wall block that was described in 2013 by Blanco et al. who presented it as an alternative to other regional anesthetic techniques. It has been described in adults as an adjunct to general anesthesia or as a primary anesthetic technique for breast surgery, it has not been widely utilized as a primary anesthetic technique in the pediatric population. It was designed to block primarily the thoracic intercostal nerves and to provide complete analgesia of the lateral part of the thorax. It provides a viable alternative to paravertebral blockade and central neuraxial block in this patient population The investigators believe that the bilateral two-level injection technique may provide effective analgesia as its efficacy was not properly investigated in corrective heart surgeries with median sternotomy in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Risk Adjustment for Congenital Heart Surgery (RACHS) category 1,2 and 3 Pediatric patients undergoing corrective congenital cardiac surgeries via a median sternotomy

Exclusion Criteria:

* Refusal of legal guardian.
* Patient with congestive heart failure .
* Patient undergoing Redo cardiac surgery.
* Known allergy to local anesthetics.
* Infection at injection site.
* Bleeding disorders (drug induced i.e., coumadin; or genetic i.e. hemophilia; or acquired i.e. DIC), coagulopathy: PTT > 40 seconds, INR > 1.4, platelet count < 100x10⁹.
* severe renal impairment (estimated Glomerular filtration rate less than 30ml/min/1.73m2) or hepatic insufficiency (Child-Pugh Class B and C).
* Neurological disorders because it will be difficult to assess their pain score (e.g. cerebral palsy).

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Fentanyl consumption | in the first 24 hours post-operatively

SECONDARY OUTCOMES:
intraoperative heart rate | Intraoperative period
  After induction of anesthesia (baseline), after skin incision, after sternotomy, during aortic cannulation, and 15 minutes after weaning from cardiopulmonary bypass
Intraoperative systolic blood pressure | Intraoperative period
  After induction of anesthesia (baseline), after skin incision, after sternotomy, during aortic cannulation, and 15 minutes after weaning from cardiopulmonary bypass
Intraoperative additional boluses of fentanyl | Intraoperative period
  additional boluses of fentanyl at a dose of 0.5 µg/kg whenever HR or SBP increased more than 20% of baseline
Postoperative heart rate | at 1, 2, 4, 8, 12, and 24 hours post-operatively
Postoperative systolic blood pressure | at 1, 2, 4, 8, 12, and 24 hours post-operatively
Postoperative FLACC score | at 1, 2, 4, 8, 12, and 24 hours post-operatively
  Postoperative pain intensity measured by "Face, Leg, Activity, Cry, Consolability" scale in children
Time to first rescue analgesia | recorded during the first 24 hours after surgery (in hours unit)
  first incidence of fentanyl bolus in the postoperative phase if FLACC score is 4 or more, targeting FLACC score of 3 or less
Time to extubation | 24 hours post-operatively
  Either within 2, 6, 12, or 24 hours after surgery
Incidence of complications | 24 hours post-operatively
  Complications including postoperative vomiting, hematoma formation, ithching, or local anesthetic toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Abu El Reesh pediatric university hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mayes J, Davison E, Panahi P, Patten D, Eljelani F, Womack J, Varma M. An anatomical evaluation of the serratus anterior plane block. Anaesthesia. 2016 Sep;71(9):1064-9. doi: 10.1111/anae.13549. Epub 2016 Jul 20. PMID 27440171
- [Background] Ren Y, Li L, Gao J, Hua L, Zheng T, Wang F, Zhang J. Regional Analgesia in Pediatric Cardiothoracic Surgery: A Bayesian Network Meta-Analysis. J Cardiothorac Vasc Anesth. 2025 Apr;39(4):1037-1048. doi: 10.1053/j.jvca.2024.12.043. Epub 2025 Jan 9. PMID 39880711
- [Background] Egbuta C, Mason KP. Current State of Analgesia and Sedation in the Pediatric Intensive Care Unit. J Clin Med. 2021 Apr 23;10(9):1847. doi: 10.3390/jcm10091847. PMID 33922824
- [Background] Mazzeffi M, Khelemsky Y. Poststernotomy pain: a clinical review. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):1163-78. doi: 10.1053/j.jvca.2011.08.001. Epub 2011 Sep 29. No abstract available. PMID 21955825
- [Background] Shenkman Z, Shir Y, Weiss YG, Bleiberg B, Gross D. The effects of cardiac surgery on early and late pulmonary functions. Acta Anaesthesiol Scand. 1997 Oct;41(9):1193-9. doi: 10.1111/j.1399-6576.1997.tb04865.x. PMID 9366943
- [Background] Sasseron AB, Figueiredo LC, Trova K, Cardoso AL, Lima NM, Olmos SC, Petrucci O. Does the pain disturb the respiratory function after open heart surgery? Rev Bras Cir Cardiovasc. 2009 Oct-Dec;24(4):490-6. doi: 10.1590/s0102-76382009000500010. English, Portuguese. PMID 20305922
- [Background] Ergun A, Sirlak M. [Pulmonary function test before and after operation of coronary artery by-pass surgery]. Tuberk Toraks. 2003;51(1):17-22. Turkish. PMID 15100899
- [Background] Zubrzycki M, Liebold A, Skrabal C, Reinelt H, Ziegler M, Perdas E, Zubrzycka M. Assessment and pathophysiology of pain in cardiac surgery. J Pain Res. 2018 Aug 24;11:1599-1611. doi: 10.2147/JPR.S162067. eCollection 2018. PMID 30197534
- [Background] Guimaraes-Pereira L, Reis P, Abelha F, Azevedo LF, Castro-Lopes JM. Persistent postoperative pain after cardiac surgery: a systematic review with meta-analysis regarding incidence and pain intensity. Pain. 2017 Oct;158(10):1869-1885. doi: 10.1097/j.pain.0000000000000997. PMID 28767509
- [Background] He Y, Xu M, Li Z, Deng L, Kang Y, Zuo Y. Safety and feasibility of ultrasound-guided serratus anterior plane block and intercostal nerve block for management of post-sternotomy pain in pediatric cardiac patients: A prospective, randomized trial. Anaesth Crit Care Pain Med. 2023 Dec;42(6):101268. doi: 10.1016/j.accpm.2023.101268. Epub 2023 Jun 24. PMID 37364851
- [Background] Kupeli I, Adilovic AS. The "Feasibility" And "Safety" Of Ultrasound Guided Bilateral Two Level Serratus Anterior Plane Block in Children With Median Sternotomy Pain: A Case Series. J Cardiothorac Vasc Anesth. 2021 Jan;35(1):270-273. doi: 10.1053/j.jvca.2020.03.020. Epub 2020 Mar 19. No abstract available. PMID 32360008
- [Background] Abdelbaser II, Mageed NA. Analgesic efficacy of ultrasound guided bilateral transversus thoracis muscle plane block in pediatric cardiac surgery: a randomized, double-blind, controlled study. J Clin Anesth. 2020 Dec;67:110002. doi: 10.1016/j.jclinane.2020.110002. Epub 2020 Jul 24. PMID 32717448
- [Background] Malviya S, Voepel-Lewis T, Burke C, Merkel S, Tait AR. The revised FLACC observational pain tool: improved reliability and validity for pain assessment in children with cognitive impairment. Paediatr Anaesth. 2006 Mar;16(3):258-65. doi: 10.1111/j.1460-9592.2005.01773.x. PMID 16490089
- [Background] Voepel-Lewis T, Zanotti J, Dammeyer JA, Merkel S. Reliability and validity of the face, legs, activity, cry, consolability behavioral tool in assessing acute pain in critically ill patients. Am J Crit Care. 2010 Jan;19(1):55-61; quiz 62. doi: 10.4037/ajcc2010624. PMID 20045849
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Tewari P, Hajela K, Ahmad SS. Bilateral superficial serratus anterior plane block in a pediatric patient for post-operative analgesia undergoing asd repair via median sternotomy- A case report. Ann Card Anaesth. 2022 Jan-Mar;25(1):116-118. doi: 10.4103/aca.aca_113_21. PMID 35075035
- [Background] Devarajan J, Balasubramanian S, Shariat AN, Bhatt HV. Regional Analgesia for Cardiac Surgery. Part 2: Peripheral Regional Analgesia for Cardiac Surgery. Semin Cardiothorac Vasc Anesth. 2021 Dec;25(4):265-279. doi: 10.1177/10892532211002382. Epub 2021 Apr 8. PMID 33827348
- [Background] Jack JM, McLellan E, Versyck B, Englesakis MF, Chin KJ. The role of serratus anterior plane and pectoral nerves blocks in cardiac surgery, thoracic surgery and trauma: a qualitative systematic review. Anaesthesia. 2020 Oct;75(10):1372-1385. doi: 10.1111/anae.15000. Epub 2020 Feb 16. PMID 32062870